CLINICAL TRIAL: NCT06737770
Title: Clinical and Functional Assessment of Patients With Transfemoral Amputation Treated With Osteointegrated Implant
Acronym: OSTEO-OUTCOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSTEO-OUTCOME
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prosthesis; Lower Limb Amputation Knee; Amputation; Traumatic, Leg, Lower
Keywords: Osseointegration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing osseointegration surgery for transfemoral amputation (Experimental)
  Interventions: Procedure: osseointegrated surgery for transfemoral amputation

INTERVENTIONS:
Procedure: osseointegrated surgery for transfemoral amputation — osseointegrated surgery for transfemoral amputation

SUMMARY:
Limb amputation is a traumatic event that significantly reduces the ability to perform daily activities, impairs mobility, and lowers quality of life. In Italy, approximately 4 million people live with disabilities, with 1.2 million having motor disabilities. Among lower limb amputees (around 200,000), most are elderly, with amputations due to diabetic or vascular issues. Other groups include middle-aged adults (often victims of workplace accidents) and young individuals (victims of traffic accidents).

Post-amputation rehabilitation mainly involves the use of prostheses, which, however, can cause skin problems due to the socket (the part that anchors the prosthesis to the residual limb). Among patients using a socket, 34-63% develop chronic skin issues and pain. Complications include excessive sweating, sores, abscesses, and irritation. Additionally, daily volume changes in the residual limb and long-term weight fluctuations further complicate the use of conventional prostheses.

In the last two decades, research groups, assisted by experienced surgeons, have worked to develop implant solutions that bypass the socket and address these issues. One such solution is osteointegrated prostheses, which use the principle of osteointegration to anchor the prosthesis directly to the bone of the residual limb. A metal stem is surgically inserted into the medullary canal of the residual limb and fixed through bone growth, establishing a direct connection between the amputated limb and the external prosthesis.

Osteointegrated prostheses are widely accepted worldwide as a valid alternative to socket prostheses, especially for young and active individuals with transfemoral, transtibial, transhumeral, or transradial amputations not caused by vascular issues. The key benefit of osteointegration is the restoration of load alignment along the anatomical and mechanical axis, improving control of the residual limb during walking, as well as overall functional capacity and quality of life. Other advantages include greater stability, enhanced sitting comfort, a wider range of hip movement, faster attachment and detachment of the prosthesis, and improved body perception. Additionally, the direct contact between the metal stem and the bone generates sensory feedback (osteoperception), allowing the patient to better control the amputated limb by perceiving ground contact through vibrations transmitted to the bone. Osteointegration offers the only viable alternative for prosthetic use in patients with a short residual limb, where conventional socket prostheses would not be suitable.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes, aged between 18 and 65 years;
* Subjects with unilateral transfemoral amputation, following trauma, tumor, infection, or congenital defect;
* Subjects already scheduled for osteointegrated prosthesis surgery for amputation;
* BMI < 35 kg/m²;
* Difficulty in using the traditional socket prosthesis (pain, reduced mobility, short residual limb, skin infections, ulcers, volume changes in the residual limb);
* Subjects who have signed informed consent and reviewed the study information sheet.

Absolute exclusion criteria:

* Peripheral vascular diseases;
* Pregnancy;
* Rheumatoid arthritis;
* Neurological deficits;
* Amputation of the contralateral limb;
* Active infections;
* Immunodeficiency;
* Comorbidities/concurrent disabilities, general or localized (Multiple Sclerosis, Parkinson's disease, muscle tone disorders, malignant neoplasms, etc.), that may interfere with the study;
* Presence of uncontrolled psychiatric comorbidities;
* Declared or evident cognitive deficits that would impair understanding of the tasks required (MMSE ≤ 24);
* Insufficient degree of cooperation;
* Length of the bone stump (measured from the lesser trochanter to the apex of the stump) less than 15 cm;
* Previous radiotherapy on the amputated limb;
* Ongoing chemotherapy treatments.

Relative exclusion criteria:

* Smoking;
* Uncontrolled diabetes;
* Previous infections;
* Presence of additional joint prostheses on the same limb;
* Osteoporosis with a T-score of -2.5 or lower.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L | 12 months after surgery
  It is a generic tool for measuring perceived quality of life in relation to health status, divided into 5 domains, each assigned a score ranging from 1 (best possible outcome) to 5 (worst possible outcome): mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Additionally, there is a domain related to general health, scored from 0 (worst possible health status) to 100 (best possible health status)

SECONDARY OUTCOMES:
Q-TFA | 12 months after surgery
  Assessment of quality of life specifically for amputee subjects through the 'Transfemoral Amputation Questionnaire' (Q-TFA), a questionnaire that evaluates prosthesis use and mobility, as well as the individual's issues and general health.
VAS | 12 months after surgery
  It is a unidimensional quantitative pain rating scale with 10 points. The scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that specific moment. 0 means no pain, and 10 indicates the worst possible pain.
ABIS | 12 months after surgery
  The Body Image Scale for Amputees is a self-administered questionnaire designed to specifically measure body image perception in amputees from the patient's perspective.
TAPES | 12 months after surgery
  The Trinity Amputation and Prosthesis Experience Scales is a self-administered questionnaire that includes the domains of psychosocial adjustment, activity restriction, and prosthesis satisfaction, each divided into 3 subscales. Additionally, it explores residual pain, phantom limb pain, and other medical issues, thus incorporating both the physical and psychosocial aspects of adaptation.
PWB-PTCQ | 12 months after surgery
  The Psychological Well-Being-Post-Traumatic Changes Questionnaire is a self-assessment tool designed to evaluate perceived changes in psychological well-being following traumatic events. The PWB-PTCQ is based on a well-established theoretical framework of psychological well-being (PWB) and adopts the general format of existing measures of growth.
WHODAS 2.0 | 12 months after surgery
  The WHO Disability Assessment Schedule is an assessment questionnaire based on the International Classification of Functioning, Disability and Health (ICF) that measures health and disability status. The questionnaire is designed to assess the level of functioning across six domains: cognitive activities, mobility, self-care, interpersonal relationships, daily living activities, and participation.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Rizzoli Orthopedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided